CLINICAL TRIAL: NCT00435253
Title: Phase 2 Study of the Biologic Lung Volume Reduction System (BLVR) in Patients With Advanced Upper Lobe Predominant Emphysema
Brief Title: US 10 mL Biologic Lung Volume Reduction (BLVR) Phase 2 Emphysema Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-C06-003
Record Dates: First submitted 2007-02-07; First posted 2007-02-14 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Pulmonary Emphysema
Keywords: emphysema; COPD; lung volume reduction; NETT; BLVR; biologic lung volume reduction; bronchoscopic lung volume reduction
MeSH Terms: conditions — Pulmonary Emphysema; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BLVR Treatment (Experimental): BLVR Treatment
  Interventions: Biological: BLVR Treatment

INTERVENTIONS:
Biological: BLVR Treatment — BLVR Treatment, 10 mL Hydrogel

SUMMARY:
Evaluate the efficacy and safety of the 10 mL BLVR System in 1 or 2 treatment sessions (8 subsegments, 4 in each lung) in patients with advanced upper lobe predominant emphysema.

DETAILED DESCRIPTION:
Prospective, open-label, non-controlled, multi-center Phase 2 Study evaluating the efficacy and safety of the 10 mL BLVR System in patients with advanced upper lobe predominant emphysema. Twenty patients will be divided into 2 groups of 10 patients each and treated under conscious sedation at a total of 8 subsegments. Group 1 will be treated in 4 subsegments in 1 lung and have a second treatment of 4 subsegments in the other lung 6 to 12 weeks later. Group 2 will receive treatment at 8 subsegments (4 in each lung) during a single treatment session if possible; if not completed in 1 session the remaining subsegments will be treated 6 to 12 weeks later. Patients will be followed 96 weeks after completion of the final BLVR treatment. All patients will receive standard medical therapy in addition to BLVR treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of advanced upper lobe predominant emphysema
* age >/= 40 years
* clinically significant dyspnea
* failure of standard medical therapy to relieve symptoms (inhaled beta agonist and inhaled anticholinergic)
* pulmonary function tests within protocol-specified ranges (post bronchodilator FEV1 < 45% predicted and experiencing < 30% or 300 mL improvement using bronchodilator; TLC > 110% predicted; RV > 150% predicted)
* 6 Minute Walk Distance >/= 150 m

Exclusion Criteria:

* alpha-1 protease inhibitor deficiency
* homogeneous disease
* tobacco use within 4 months of initial visit
* body mass index < 15 kg/m2 or > 35 kg/m2
* clinically significant asthma, chronic bronchitis or bronchiectasis
* allergy or sensitivity to procedural components
* pregnant, lactating or unwilling to use birth control if required
* prior lung volume reduction surgery, lobectomy, pneumonectomy, lung transplant, endobronchial valve placement, airway stent placement or pleurodesis
* comorbid condition that could adversely influence outcomes
* inability to tolerate bronchoscopy under conscious sedation (or anesthesia)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Reduction in gas trapping | 12 weeks post treatment
SAEs - Safety of treatment and the procedure | 2 years

SECONDARY OUTCOMES:
Improvement in vital capacity | 12 weeks post treatment
Improvement in expiratory flow | 12 weeks post treatment
Improvement in inspiratory flow | 12 weeks post treatment
Improvement in dyspnea symptoms (breathlessness) | 12 weeks post treatment
Improvement in exercise capacity | 12 weeks post treatment
Improvement in respiratory quality of life | 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Victor Pinto-Plata, MD, Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.; Gerard Criner, MD, Principal Investigator — Temple University Lung Center; Mark Gotfried, MD, Principal Investigator — Pulmonary Associates; Charlie Strange, MD, Principal Investigator — Medical Univ South Carolina Hospital; Mark Dransfield, MD, Principal Investigator — Univ of Alabama Birmingham Lung Health Center
Locations (5):
- United States (5):
  - University of Alabama Birmingham Lung Health Center, Birmingham, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - Caritas St Elizabeth's Med Cen, Boston, Massachusetts
  - Temple University Lung Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina Hospital, Charleston, South Carolina

REFERENCES:
- [Background] Ingenito EP, Berger RL, Henderson AC, Reilly JJ, Tsai L, Hoffman A. Bronchoscopic lung volume reduction using tissue engineering principles. Am J Respir Crit Care Med. 2003 Mar 1;167(5):771-8. doi: 10.1164/rccm.200208-842OC. Epub 2002 Oct 11. PMID 12406835
- [Background] Reilly J, Washko G, Pinto-Plata V, Velez E, Kenney L, Berger R, Celli B. Biological lung volume reduction: a new bronchoscopic therapy for advanced emphysema. Chest. 2007 Apr;131(4):1108-13. doi: 10.1378/chest.06-1754. PMID 17426216
- [Derived] Criner GJ, Pinto-Plata V, Strange C, Dransfield M, Gotfried M, Leeds W, McLennan G, Refaely Y, Tewari S, Krasna M, Celli B. Biologic lung volume reduction in advanced upper lobe emphysema: phase 2 results. Am J Respir Crit Care Med. 2009 May 1;179(9):791-8. doi: 10.1164/rccm.200810-1639OC. Epub 2009 Jan 29. PMID 19179484